CLINICAL TRIAL: NCT06712030
Title: Effect of Pharmacological Treatment with Angiotensin Receptor/Neprilysin Inhibitors on Transthyretin Cardiac Amyloidosis and Heart Failure with Reduced Ejection Fraction (SAVA-TTR)
Brief Title: Effect of Angiotensin Receptor/Neprilysin Inhibitors on Transthyretin Cardiac Amyloidosis and Heart Failure with Reduced Ejection Fraction
Acronym: SAVA-TTR
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Esther Gonzalez López, Principal Investigator, Puerta de Hierro University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-515661-34-00; 2024-515661-34-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-19; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Transthyretin Amyloidosis Cardiomyopathy (ATTR-CM)
Keywords: Heart failure; Reduced ejection fraction; Angiotensin receptor/neprilysin inhibitors; Sacubitril valsartan
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The analysis of the echocardiogram will be performed by evaluators blinded to the treatment and the timing of the imaging.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sacubitril/Valsartan (Experimental): Sacubitril/valsartan up to maximum tolerated dose
  Interventions: Drug: Sacubitril / Valsartan
- No treatment (No Intervention): No initiation of Sacubitril/valsartan

INTERVENTIONS:
Drug: Sacubitril / Valsartan — Dose titration of Sacubitril/Valsartán to the maximum tolerated dose (maximum 97/103 mg)
  Arms: Sacubitril/Valsartan

SUMMARY:
Prospective, randomized, multicenter, open-label clinical trial to evaluate the safety and efficacy of Sacubitril/Valsartan (Sac/Vals) compared to no initiation of the drug in patients with transthyretin cardiac amyloidosis (ATTR) and heart failure with reduced ejection fraction (LVEF ≤40%). The primary objective is to determine the impact of Sac/Vals treatment on systolic function by assessing the change in LVEF on echocardiogram at 12-month follow-up.

DETAILED DESCRIPTION:
Transthyretin cardiac amyloidosis (ATTR) has emerged as a prevalent and underdiagnosed cause of heart failure (HF), affecting patients both with preserved left ventricular ejection fraction (LVEF) and with systolic dysfunction. It remains unclear whether this population benefits from standard treatments for HF with reduced LVEF or whether treatment with renin-angiotensin system inhibitors and neprilysin might even be harmful in ATTR.

The investigators plan to conduct a prospective, randomized, multicenter, open-label clinical trial to evaluate the safety and efficacy of Sacubitril/Valsartan (Sac/Vals), as recommended in current HF guidelines, versus no treatment in patients with ATTR and heart failure with reduced ejection fraction (HFrEF), including those with LVEF ≤40%.

Approximately 114 patients from four Spanish centers will be randomized 1:1 to receive Sac/Vals treatment (up to the maximum tolerated dose) or to not initiate the drug, with stratification by center and tafamidis treatment. It has been included a run-in period with a low dose of Sac/Vals to assess tolerance prior to randomization. Patients will have scheduled follow-up visits at 3, 6, and 12 months, during which clinical, functional, analytical, electrocardiographic, and echocardiographic variables will be evaluated.

The primary objective is to determine the impact of Sac/Vals treatment on systolic function in patients with ATTR and HFrEF by assessing the change in LVEF on echocardiogram at 12 months. Improvement in LVEF will be defined as an increase of ≥5% from the baseline echocardiogram to the 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age of both sexes.
* Patients diagnosed with ATTR cardiac amyloidosis as indicated in guidelines, both in its hereditary form (ATTRv) or wild-type form (ATTRwt).
* Patients initially evaluated or under follow-up in Cardiomyopathy/Heart Failure/Amyloidosis Units at participating centers.
* Heart failure and reduced ejection fraction: LVEF ≤40%, in functional class I, II, or III according to the New York Heart Association (NYHA).

Exclusion Criteria:

* NYHA Functional Class IV.
* Stage 4 and 5 chronic kidney disease (creatinine clearance by CKD-EPI <30 mL/min/1.73m²).
* Hyperkalemia (blood potassium levels > 5.4 mmol/L).
* Hypotension defined as systolic blood pressure (SBP) <100 mmHg on two consecutive measurements.
* Treatment with ACE inhibitors, ARBs, or sacubitril/valsartan at the time of enrollment.
* History of angioedema or hypersensitivity to ACE inhibitors or ARBs.
* Treatment with TTR gene silencers or diflunisal.
* Participation in another clinical trial.
* Pregnancy, breastfeeding, or fertile women unwilling to use adequate contraception throughout the study duration.
* Any condition that, in the investigator's opinion, compromises participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular systolic function (%) assessed by echocardiogram. | 12 months
  Measured by biplane method in percentage

SECONDARY OUTCOMES:
Change in left ventricular systolic function assessed by global longitudinal strain (GLS) | 12 months
  Measure of longitudinal shortening as a percentage
Change in E/e' ratio measured by echocardiogram. | 12 months
  Ratio between E wave (peak velocity of early diastolic blood flow across the mitral valve, measured using transmitral Doppler) and E' (E prime): velocity of early diastolic mitral annular motion, measured using tissue Doppler imaging.
Change in functional capacity assessed by 6-minute walk test | 12 months
  Distance covered over a time of 6 minutes in a flat surface in meters.
Change in quality of life according to the Kansas City Cardiomyopathy Questionnaire | 12 months
  0 to 100 scale, where 0 is the worst possible health status and 100 best possible health status.
Change in N-terminal pro-B-type natriuretic peptide (NTproBNP) biomarker level. | 12 months
  Measure in blood. Unit pg/ml.
Proportion of patients experiencing cardiovascular hospitalizations. | 12 months
Proportion of patients experiencing adverse events | 12 months
  Including serious adverse event, grade 3-4 adverse event, adverse reaction, adverse event of special interest.
Proportion of patients discontinuing treatment | 12 months
Proportion of patients experiencing all-cause mortality. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Esther Gonzalez Lopez, MD, PhD, Principal Investigator — Heart Failure and Inherited Cardiac Diseases Unit, Department of Cardiology, Hospital Universitario Puerta de Hierro, IDIPHISA, Madrid, Spain
Locations (1):
- Hospital Universitario Puerta de Hierro, Majadahonda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Under agreement, individual or aggregated patient data could be shared with other scientific groups for scientific projects. Data can be shared only for scientific purposes and in full compliance with Personal Data Protection requirements in the EU.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After study scientific publication
Access Criteria: Under request to Study Chair